CLINICAL TRIAL: NCT05685108
Title: Optimizing Ultrasound-induced Anti-inflammation in Human Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mark Okusa, MD, Chief, Division of Nephrology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSR220029
Record Dates: First submitted 2022-12-15; First posted 2023-01-13 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects
Keywords: Cholinergic anti-inflammatory pathway; Vagus nerve; Cytokines; Neuromodulation

STUDY DESIGN:
Intervention Model Description: After screening, eligible participants will be assigned to one of the two groups and randomized to order of treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1 (Active Comparator): In Subgroup 1, individuals will receive pulsed ultrasound with a mechanical index of 0.6 and 1.4 delivered to the splenic hilum.
  In Subgroup 2, individuals will receive pulsed ultrasound with a mechanical index of 1.0 and 1.8 delivered to the splenic hilum.
  In Subgroup 3, individuals will receive sham treatment and pulsed ultrasound with a mechanical index of 1.4 delivered to the splenic hilum.
  In all Subgroups, the two doses will be administered in separate visits with min. 14 days between each stimulation.
  Interventions: Device: Ultrasound stimulation intensity
- Group 2 (Active Comparator): Individuals will receive pulsed ultrasound with a mechanical index of 1.4 delivered to the splenic hilum and the cervical vagus nerve. The two doses will be administered in separate visits with min. 14 days between each stimulation.
  Interventions: Device: Ultrasound stimulation site

INTERVENTIONS:
Device: Ultrasound stimulation intensity — A clinical ultrasound transducer will be placed against the abdomen or neck of an individual in order to administer insonification to the splenic nerve.
  Arms: Group 1
Device: Ultrasound stimulation site — A clinical ultrasound transducer will be placed against the abdomen or neck of an individual in order to administer insonification to the splenic nerve and the cervical vagus nerve.
  Arms: Group 2

SUMMARY:
This is a feasibility study to determine whether pulsed ultrasound stimulation targeting the splenic nerve or the cervical vagus nerve can elicit an anti-inflammatory immune response in healthy volunteers.

DETAILED DESCRIPTION:
Recent advances have shown that neural pathways are able to regulate immunity and inflammation. The cholinergic anti-inflammatory pathway is a well-characterized neural circuit that consists of the vagus nerve to spleen circuit, which has been stimulated with implantable devices to improve autoimmune conditions such as rheumatoid arthritis.

Recently, the use of pulsed ultrasonic waves to modulate the neuroimmune pathway has gained interest due to its potential in treating inflammatory disorders non-invasively. This study is designed to test the hypothesis that pulsed ultrasound stimulation can be used effectively in human subjects to control pathogenic inflammatory responses. The overall goal of this project is to determine which, if any, ultrasound stimulation protocols are able to restrict the inflammatory response of immune cells collected from healthy subjects post-ultrasound stimulation.

Four different levels of ultrasound intensity ("doses") will be tested in this study to determine the dose(s) capable of producing an anti-inflammatory effect. The doses will be defined in terms of mechanical index and each subject will receive two different doses of ultrasound. In addition, the study will investigate the efficacy of cervical vagus (neck)-targeted ultrasound, given that it may have an effect similar to spleen-targeted ultrasound through upstream vagus nerve modulation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 25-50 years
* Provision of signed and dated informed consent form
* Able to comprehend the study goals and procedures, stated willingness to comply with all study procedures, and availability for the duration of the study
* Considered English proficient so that the subject can follow verbal commands during the ultrasound procedure
* In good general health, as evidenced by medical history
* Laboratory results indicating normal blood count and adequate organ function
* Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

* Chronic medical conditions, including cancer (in remission or active cancer), cerebrovascular disease, chronic kidney disease, heart conditions (such as heart failure, coronary artery disease, cardiomyopathies), lung disease, liver disease, hypertension, diabetes mellitus type 1 and 2, human immunodeficiency virus infection, primary immunodeficiencies, solid organ or hematopoietic cell transplantation, tuberculosis, and cystic fibrosis, autoimmune disorders (e.g., rheumatoid arthritis, inflammatory bowel disease), sickle cell anemia or other anemia syndromes
* Mean systolic and diastolic blood pressure values during screening of ≥160 and ≥100 mm Hg, respectively, hypertension on non-selective beta-blockers and/or alpha-methyl dopa, or hypertension requiring more than two anti-hypertension medications
* Obesity (body mass index ≥30 kg/m2)
* Use of anti-inflammatory or immunomodulatory medication, such as non- steroidal anti-inflammatory drugs (NSAIDs), corticosteroids, or other immunosuppressants, within one week of receiving ultrasound delivery
* Use of anticoagulant drugs (e.g., coumadin, direct oral anticoagulants) or antiplatelet drugs (e.g., aspirin, clopidogrel) within one week of receiving ultrasound delivery
* Pregnancy, breastfeeding, or planning to become pregnant during the study
* Active bacterial or viral infection; febrile illness within 2 weeks of receiving ultrasound delivery
* Known allergic reactions to ultrasound gel
* Treatment with another investigational drug or other intervention within 1 month of receiving ultrasound delivery
* Any vaccination received within 1 month of receiving ultrasound delivery
* Current smoker or nicotine use within 2 weeks of receiving ultrasound delivery
* Use of recreational drugs within 2 weeks of receiving ultrasound delivery
* History of arrythmia (e.g., clinically significant bradycardia, atrial flutter, atrial fibrillation, ventricular arrythmias)
* History of deep vein thrombosis or pulmonary embolism
* History of bleeding disorder
* History of seizure
* History of unilateral or bilateral vagotomy
* Participants with an implantable medical device, such as pacemaker, hearing aid implant, or any implanted electronic device
* Surgery or traumatic injury (e.g., visceral injury, cerebral injury) in the past 3 months
* Prior surgery on thyroid or parathyroid glands, esophagus, stomach, or spleen
* Participant is considered by the Investigator, after reviewing medical and psychiatric history, physical examination, and laboratory evaluations, to be unsuitable for any other reason that may either place the patient at increased risk during participation or interfere with the interpretation of the study. outcomes.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in concentrations of immune cells and cytokines depending on ultrasound stimulation intensity | Immune cells will be stimulated and assessed prior to and within 24 to 48 hours post-ultrasound treatment. Results of Luminex analysis of the pre- and post-ultrasound stimulation supernatants will be compared to quantify the impacts of the treatment.
  The primary outcome is to determine ultrasound intensities that have a biological effect on immune cells measured as a statistically significant change in the level of cytokines produced by immune cells. White blood cells will be isolated from peripheral blood and treated ex vivo with inflammatory stimuli to evaluate their capacity for cytokine production. The cytokines to be measured are (all will be measured in pg/ml): sCD40L; EGF; Eotaxin; FGF-2; FLT-3L; Fractalkine; G-CSF; GM-CSF; GRO; IFNα2; IFNy; IL-1α; IL-1β; IL-1Ra; IL-2; IL-3; IL-4; IL-5; IL-6; IL-7; IL-8; IL-9; IL-10; IL-12p40; IL-12p70; IL-13; IL-15; IL-17A; IL-17E; IL-17F; IL-18; IL-22; IL-27; IP-10; MCP-1; MCP-3; M-CSF; MDC; MIG; MIP-1α; MIP-1β; PDGF-AA; PDGF-AB/BB; TGFα; TNFα; TNFβ; VEGF-A.
Change in concentrations of immune cells and cytokines depending on ultrasound stimulation site | Immune cells will be stimulated and assessed prior to and within 24 to 48 hours post-ultrasound treatment. Results of Luminex analysis of the pre- and post-ultrasound stimulation supernatants will be compared to quantify the impacts of the treatment.
  The primary outcome is to determine the effects of spleen-targeted versus cervical vagus-targeted ultrasound stimulation on the inflammatory capacity of immune cells. This will be measured by stimulating white blood cells from peripheral blood ex vivo with inflammatory stimuli to evaluate their capacity for cytokine production. The cytokines to be measured are (all will be measured in pg/ml): sCD40L; EGF; Eotaxin; FGF-2; FLT-3L; Fractalkine; G-CSF; GM-CSF; GRO; IFNα2; IFNy; IL-1α; IL-1β; IL-1Ra; IL-2; IL-3; IL-4; IL-5; IL-6; IL-7; IL-8; IL-9; IL-10; IL-12p40; IL-12p70; IL-13; IL-15; IL-17A; IL-17E; IL-17F; IL-18; IL-22; IL-27; IP-10; MCP-1; MCP-3; M-CSF; MDC; MIG; MIP-1α; MIP-1β; PDGF-AA; PDGF-AB/BB; TGFα; TNFα; TNFβ; VEGF-A.

SECONDARY OUTCOMES:
Distribution of immune cells | The secondary outcome will be assessed before and max 48-hours after receiving ultrasound stimulation.
  The secondary outcome is to determine the effects of ultrasound stimulation on the distribution of immune cells measured as a statistically significant change in the distribution of white blood cells using flow cytometry associated with the inflammatory response following delivery of ultrasound.

OTHER OUTCOMES:
Participant comfort, experience, and new-onset sensations by questionnaire | The outcome will be assessed immediately after, within 24 to 48 hours, and 2 weeks after receiving ultrasound stimulation
  Participants will complete a questionnaire based on a dichotomous scale ("yes" or "no") to evaluate their experience of discomfort and new-onset sensations following ultrasound stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Okusa, MD, FASN, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Division of Nephrology; Center for Immunity, Inflammation & Regenerative Medicine, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there are no plans to make individual participant data available.

REFERENCES:
- [Background] Okusa MD, Rosin DL, Tracey KJ. Targeting neural reflex circuits in immunity to treat kidney disease. Nat Rev Nephrol. 2017 Nov;13(11):669-680. doi: 10.1038/nrneph.2017.132. Epub 2017 Oct 3. PMID 28970585
- [Background] Cai J, Nash WT, Okusa MD. Ultrasound for the treatment of acute kidney injury and other inflammatory conditions: a promising path toward noninvasive neuroimmune regulation. Am J Physiol Renal Physiol. 2020 Jul 1;319(1):F125-F138. doi: 10.1152/ajprenal.00145.2020. Epub 2020 Jun 8. PMID 32508112
- [Background] Gigliotti JC, Huang L, Bajwa A, Ye H, Mace EH, Hossack JA, Kalantari K, Inoue T, Rosin DL, Okusa MD. Ultrasound Modulates the Splenic Neuroimmune Axis in Attenuating AKI. J Am Soc Nephrol. 2015 Oct;26(10):2470-81. doi: 10.1681/ASN.2014080769. Epub 2015 Feb 2. PMID 25644106
- [Background] Cotero V, Fan Y, Tsaava T, Kressel AM, Hancu I, Fitzgerald P, Wallace K, Kaanumalle S, Graf J, Rigby W, Kao TJ, Roberts J, Bhushan C, Joel S, Coleman TR, Zanos S, Tracey KJ, Ashe J, Chavan SS, Puleo C. Noninvasive sub-organ ultrasound stimulation for targeted neuromodulation. Nat Commun. 2019 Mar 12;10(1):952. doi: 10.1038/s41467-019-08750-9. PMID 30862827

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT05685108/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT05685108/ICF_001.pdf